CLINICAL TRIAL: NCT03063645
Title: A Phase 1, Pilot, Single-Dose, 3-Way Crossover Study to Compare the Pharmacokinetics of AC 1202 and Two Doses of AC-SD-01 on Ketone Body Production
Brief Title: Study to Compare the Pharmacokinetics of AC 1202 and Two Doses of AC-SD-01 on Ketone Body Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-17-014_BE
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: Healthy volunteer; AC-1202; AC-SD-01; Pharacokinetic; ketone body
MeSH Terms: interventions — AC-1202

STUDY DESIGN:
Intervention Model Description: 16 healthy subjects enrolled, each subject will receive 1 dose of each treatment, with a 2 day washout in between.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group ABC (Experimental): AC-1202, AC-SD-01 (50g), AC-SD-01 (75g)
  Interventions: Drug: AC-1202; Drug: AC-SD-01 (50 g); Drug: AC-SD-01 (75 g)
- Group BCA (Experimental): AC-SD-01 (50g), AC-SD-01 (75g), AC-1202
  Interventions: Drug: AC-1202; Drug: AC-SD-01 (50 g); Drug: AC-SD-01 (75 g)
- Group CAB (Experimental): AC-SD-01 (75g), AC-1202, AC-SD-01 (50g)
  Interventions: Drug: AC-1202; Drug: AC-SD-01 (50 g); Drug: AC-SD-01 (75 g)

INTERVENTIONS:
Drug: AC-1202 — 60 g AC-1202 mixed in 240 mL of water at Hour 0 Day 1
Drug: AC-SD-01 (50 g) — 50 g AC-SD-01 mixed in 240 mL of water at Hour 0 Day 1
Drug: AC-SD-01 (75 g) — 75 g AC-SD-01 mixed in 240 mL of water at Hour 0 Day 1

SUMMARY:
To compare serum ketone body (i.e., total ketones, β hydroxybutyrate, and estimate of acetoacetate) levels after single dose administration of AC-1202 and 2 doses of AC-SD-01.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male 19-55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to Day -1 of Period 1 and throughout the study.
3. Body mass index (BMI) ≥ 20.0 and ≤ 30.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee. At screening, subjects must have alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) < the upper limit of normal and triglyceride levels must be < 250 mg/dL.
5. A non vasectomized subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to Day -1 of Period 1. A subject who has been vasectomized less than 4 months prior to Day -1 of Period 1 must follow the same restrictions as a non vasectomized male).
6. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to Day -1 of Period 1.
5. History or presence of galactosemia or hypersensitivity or idiosyncratic reaction to the study drugs, related compounds, milk, palm or coconut oil, or soy.
6. History or presence of diverticular disease, ulcers, inflammatory bowel disease or recurrent diarrhea or gout.
7. Positive urine drug or alcohol results at screening or check in.
8. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
9. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
10. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
11. QTcF interval is > 460 msec or subject has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
12. Estimated creatinine clearance ≤ 80 mL/min at screening.
13. Unable to refrain from or anticipates the use of any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to Day -1 of Period 1 and throughout the study. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study.
14. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 28 days prior to Day -1 of Period 1 and throughout the study.
15. Is lactose intolerant.
16. Is unable to complete the meal prior to Hour 0 on Day -1 of Period 1 and prior to dosing on Day 1 of Period 1.
17. Subject consumed grapefruit or Seville oranges within 14 days prior to Day -1 of Period 1.
18. Donation of blood or significant blood loss within 56 days prior to Day -1 of Period 1.
19. Plasma donation within 7 days prior to Day -1 of Period 1.
20. Participation in another clinical study within 28 days prior to Day -1 of Period 1. The 28 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day -1 of Period 1 of the current study.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-11 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
total ketones AUC0-t | 0-24 hrs
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
total ketones AUC0-inf | 0-24 hrs
  The area under the concentration-time curve from time 0 extrapolated to infinity. AUC0-inf is calculated as the sum of AUC0-t plus the ratio of the last measurable serum concentration to the elimination rate constant.
total ketones AUC%extap | 0-24 hrs
  Percent of AUC0-inf extrapolated, represented as (1 - AUC0-t/AUC0-inf)*100
total ketones Cmax | 0-24 hrs
  Maximum observed concentration
total ketones Kel | 0-24 hrs
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., there or more non-zero serum concentrations)
total ketones T 1/2 | 0-24 hrs
  Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel
total ketones Tmax | 0-24 hrs
  Time to reach Cmax. If the value occurs at more than one time points, Tmax is defined as the first time point with this value
β hydroxybutyrate AUC0-t | 0-24 hrs
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
β hydroxybutyrate AUC0-inf | 0-24 hrs
  The area under the concentration time curve from time 0 extrapolated to infinity. AUC0inf is calculated as the sum of AUC0t plus the ratio of the last measurable serum concentration to the elimination rate constant.
β hydroxybutyrate AUC%extap | 0-24 hrs
  Percent of AUC0-inf extrapolated, represented as (1 AUC0t/ AUC0inf)* 100
β hydroxybutyrate Cmax | 0-24 hrs
  Maximum observed concentration
β hydroxybutyrate Kel | 0-24 hrs
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more nonzero serum concentrations)
β hydroxybutyrate T 1/2 | 0-24 hrs
  Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel
β hydroxybutyrate Tmax | 0-24 hrs
  Time to reach Cmax. If the value occurs at more than one time point, Tmax is defined as the first time point with this value
estimate of acetoacetate AUC0-t | 0-24 hrs
  Difference between total ketones AUC0-t and total β hydroxybutyrate AUC0-t
estimate of acetoacetate AUC0-inf | 0-24 hrs
  Difference between total ketones AUC0-inf and total β hydroxybutyrate AUC0-inf
estimate of acetoacetate AUC%extap | 0-24 hrs
  Difference between total ketones AUC%extap and total β hydroxybutyrate AUC%extap
estimate of acetoacetate Cmax | 0-24 hrs
  Difference between total ketones Cmax and total β hydroxybutyrate Cmax
estimate of acetoacetate Kel | 0-24 hrs
  Difference between total ketones Kel and total β hydroxybutyrate Kel
estimate of acetoacetate T 1/2 | 0-24 hrs
  Difference between total ketones T 1/2 and total β hydroxybutyrate T 1/2
estimate of acetoacetate Tmax | 0-24 hrs
  Difference between total ketones Tmax and total β hydroxybutyrate Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tomek, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No